CLINICAL TRIAL: NCT01393925
Title: Effect of Parecoxib on Postoperative Shoulder Pain After Gynecological Laparoscopy.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Xuyu Zhang, Attending doctor, First Affiliated Hospital, Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FirstSunYetSen
Record Dates: First submitted 2011-07-11; First posted 2011-07-13 (Estimated); Last update posted 2011-11-22 (Estimated); Status verified 2011-11

CONDITIONS: Anti-Inflammatory Agents, Non-Steroidal; Pain, Postoperative; Laparoscopy
MeSH Terms: conditions — Pain, Postoperative | interventions — parecoxib

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- parecoxib, normal saline (Experimental)
  Interventions: Drug: parecoxib

INTERVENTIONS:
Drug: parecoxib — parecoxib 40mg at 30min before the end of surgery, at 8h and 20h after the surgery, intravenously

SUMMARY:
This prospective, double blind, placebo-controlled, parallel group study will be conducted in the first affiliated hospital of Sun yat-sen university in Guangzhou, China. Patients aged 18-65 (ASA I-II) undergoing elective gynecologic laparoscopic surgery with general anesthesia will be involved in this study. According to previous studies and our pilot trial, the sample size was estimated to be 120 subjects. All eligible patients will be randomly assigned to one of three groups: Group A (single parecoxib) receiving parecoxib 40mg at 30min before the end of surgery; Group B (multiple parecoxib) receiving parecoxib 40mg at 30min before the end of surgery, at 8h and 20h after the surgery, respectively, and Group C (Control group) receiving normal saline. All patients will be managed by a standard propofol-remifentanil based total intravenous anesthesia protocol. The incidence and intensity of shoulder pain at rest and with motion will be evaluated by an independent doctor blinding to medication and grouping using visual analog scale (VAS) at 6h, 24h and 48h postoperatively. Other types of pain (e.g. trocar wound and visceral pain), side effects (such as postoperative nausea and vomiting, itching, dizziness, and oversedation) will be assessed as well. At the end of the observation, the intensity of the maximum pain will be recorded, and the effect of shoulder pain on the four variables regarding to quality of life (activity, mood, walking and sleep) will be assessed using modified Brief Pain Inventory(BPI) questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* females age 18-65yr
* American Society of Anesthesiologists (ASA) physical status classification I-II
* Body Mass Index(BMI) 18-25kg/m2
* scheduled for elective gynecologic laparoscopic surgery

Exclusion Criteria:

* patients with a history of severe cardiac, pulmonary, hepatic, renal disease, chronic drug or alcohol abuse;
* the presence of preoperative shoulder pain or any chronic pain syndrome, long-term use of analgesics;
* allergy or contraindications to nonsteroidal anti-inflammatory drugs (allergy, peptic ulcer disease, gastroesophageal reflux disease, renal insufficiency, coagulopathy) and any other drugs used in the study;
* those whose pain evaluation was judged unreliable

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2011-07; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
The incidence of shoulder pain | up to 15 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology,,The first affiliated hospital of Sun Yat-Sen university, Guangzhou, Guangdong, China